CLINICAL TRIAL: NCT02051491
Title: A Randomized Controlled Trial of BiPhasic Nasal Continuous Positive Airway Pressure (BP-NCPAP) vs. Non-invasive High Frequency Ventilation (NIHFV) Following NCPAP Failure: A Pilot Study
Brief Title: Non-invasive Ventilation for Extubation Success in Infants Less Than 1,250 Grams
Acronym: NOVEL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Principal Investigator, Vibhuti Shah, Staff Neonatologist, Mount Sinai Hospital, Mount Sinai Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-0276A
Record Dates: First submitted 2013-11-08; First posted 2014-01-31 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-05

CONDITIONS: Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BP-NCPAP (Active Comparator): Nasal BP-NCPAP will be delivered using the Infant Flow® SiPAP™ and either nasal prongs or mask interface. A blood gas (arterial if an arterial line exists, or a capillary sample) will be drawn at the time of NCPAP failure (time 0) unless one was done within 1 hour preceding the randomization. The blood gas will then be repeated at 1 hour and recorded along with transcutaneous carbon dioxide (TcCO2) monitor data (if available). Initial settings of BP-NCPAP will be a lower level PEEP of 5 cm water (H2O) and a higher level PEEP of 8 cm H2O at a cycle rate of 20 per minute with 1 second at the higher PEEP per cycle. The settings can then be adjusted and titrated up to a maximum of 7 and 10 cm H2O for the lower and higher PEEPs respectively at a maximum rate of 30 cycles per second based on fraction of inspired oxygen (FiO2) requirements.
  Interventions: Device: BP-NCPAP
- NIHFV (Experimental): NIHFV will be provided using the Drager VN500, using either nasal prong or mask interfaces.A blood gas (arterial if an arterial line exists, or a capillary sample) will be drawn at the time of NCPAP failure (time 0) unless one was done within 1 hour preceding the randomization. The blood gas will then be repeated at 1 hour and recorded along with TcCO2 monitor data (if available). Initial settings for NIHFV arm will be MAP of 8 cm H2O, frequency of 10 Hz, and amplitude of 20 cm H2O. The maximum allowable MAP will be 10 cm of H2O. The range of frequency allowed will be 6 - 14 Hz. Both frequency and amplitude will be adjusted to try and achieve palpable/visible chest movement and to achieve target CO2 levels for the particular patient.
  Interventions: Device: NIHFV

INTERVENTIONS:
Device: BP-NCPAP — Initial settings of BP-NCPAP will be a lower level PEEP of 5 cm H2O and a higher level PEEP of 8 cm H2O at a cycle rate of 20 per minute with 1 second at the higher PEEP per cycle. The settings can then be adjusted and titrated up to a maximum of 7 and 10 cm H2O for the lower and higher PEEPs respectively at a maximum rate of 30 cycles per second based on FiO2 requirements.
  Other Names: InfantFlow® SiPAP™
  Arms: BP-NCPAP
Device: NIHFV — The initial settings will be a MAP of 8 cm H2O, frequency of 10 Hz, and amplitude of 20 cm H2O. The maximum allowable MAP will be 10 cm of H2O. The range of frequency allowed will be 6 - 14 Hz. Both frequency and amplitude will be adjusted to try and achieve palpable/visible chest movement and to achieve target CO2 levels for the particular patient.
  Other Names: Drager VN500
  Arms: NIHFV

SUMMARY:
In preterm infants, endotracheal mechanical ventilation is well known to cause various forms of lung injury including volutrauma, barotrauma and oxytrauma - collectively known as ventilator-induced lung injury (VILI). As such, there is a move towards non-invasive ventilation (NIV) in recent decades. However, many infants placed on NIV modes fail and require intubation. A relatively recent mode of NIV is non-invasive high frequency ventilation (NIHFV). Studies on this modality are scarce, but do suggest that neonates can be ventilated effectively. However, its efficacy in comparison with other existing modes of NIV remains unknown due to lack of appropriate studies. The investigators hypothesize that NIHFV is a superior NIV mode than Biphasic Nasal Continuous Positive Airway Pressure (BP-NCPAP) in preterm infants in preventing intubation following NCPAP failure.

DETAILED DESCRIPTION:
Intubation and mechanical ventilation has long been the mainstay in managing infants with respiratory disease in the neonatal intensive care unit (NICU). However, in recent decades, the use of endotracheal mechanical ventilation (EMV) has been implicated as a major cause of ventilator-induced lung injury (VILI).Prolonged endotracheal intubation in the neonate has been linked with morbidities including bronchopulmonary dysplasia (BPD), nosocomial pneumonia, air leak syndromes and subglottic stenosis. Moreover, BPD has been linked with impaired neurodevelopmental outcome.

There has been a conscious effort amongst neonatologists to reduce the duration of EMV to minimize these undesirable side effects. Non-invasive ventilatory support has been increasingly used to that effect in recent years. Various forms of NIV including NCPAP, BP-NCPAP and nasal intermittent positive pressure ventilation (NIPPV) have become part of the ventilatory management of neonates in NICUs across the globe.

Originally described in the early 1970s,9 the use NCPAP has seen renewed interest since the 1990s when the significance of VILI became apparent. In retrospective studies, NCPAP has been shown to reduce the rates of bronchopulmonary dysplasia (BPD). A recent multi-center prospective randomized controlled trial of infants between 25 and 28 week gestation showed that infants treated with early NCPAP required fewer days of ventilation and had a reduced oxygen dependency after 28 days (although not at 36 weeks corrected GA). A subsequent analysis of these patients showed improved lung mechanics and gas exchange. However NCPAP use is not without its risks. Air leak syndromes, diminished cardiac output, gaseous distention and nasal injury/excoriations are well described complications of its use. Despite these drawbacks, NCPAP remains an efficacious modality to help reduce endotracheal intubation and limit VILI.

Although successful in reducing the reliance on EMV, it is also well known that up to 43-80% of neonates with moderate to severe respiratory disease treated with NCPAP fail and require intubation. BiPhasic NCPAP and NIPPV have been used with increasing frequency in NICUs in recent years to help prevent re-intubation, but with limited evidence guiding their use.

BiPhasic-NCPAP, described in the late 1980s as a form of augmented ventilation, provides two levels of non-invasive pressure support, typically cycled between 20-30 times per minute and the upper level of support usually lasting one second. As in NCPAP, the patient breathes around the two levels of pressures provided. However, there is currently no evidence to suggest that the use of BP-NCPAP offers any advantage over NCPAP. In a recent randomized controlled prospective study from the investigators centre comparing BP-NCPAP (N=69) and NCPAP (N=67), the former was not shown to be superior to the latter in facilitating sustained extubation in infants < 1,250 grams (67% vs. 58%, P = 0.27). Nevertheless, it is presumed that BP-NCPAP offers the same benefits as NCPAP, and remains in use as a rescue mode of NIV across many NICUs after NCPAP failure.

NIPPV is yet another NIV mode, offering a combination of NCPAP superimposed with ventilator provided peak inspiratory pressure (PIP) via a non-invasive interface, designed to mimic and augment the spontaneous breathing of neonates as in EMV. The PIP provided can be both synchronized or non-synchronized with patient breaths. However there is potential for significant inaccuracies in the synchronization process. Furthermore, the Infant Star ventilator with the Graseby capsule, one of the prototype ventilators capable of providing synchronized NIPPV, is no longer available. Despite this limitation, NIPPV remains in use in both non-synchronized and synchronized forms.8 At this time, to the best of the investigators knowledge, no studies have compared BP-NCPAP and NIPPV directly. In fact, in the recently completed NIPPV trial by Kirpalani et al BP-NCPAP and NIPPV were included in the same arm, which failed to show a reduction in the incidence of BPD compared to the NCPAP arm.

Based on studies conducted so far there is no firm consensus on what is the best non-invasive mode to be used and the modality of choice remains an individual decision depending on the preference and experience of the specific unit. Noninvasive high frequency ventilation is an alternative and relatively new mode of NIV and has been explored in 4 clinical studies so far (appendix A). In a study of 21 preterm and term infants, patients were switched from NCPAP to NIHFV to promote carbon dioxide (CO2) elimination and continued for a mean of 35 (2-144) hours. The authors reported that the partial pressure of carbon dioxide (PaCO2) decreased with the use of this modality from 8.3 to 7.2 kilo pascal (KPa). The major limitations of this study include the heterogeneity of patient population, the etiologies of primary lung disease, small sample size and lack of any control group. In a more recent study by Colaizy et al, NIHFV was used in 14 subjects for a period of 2 hours and a trend towards a decrease in PaCO2 levels was noted with the use of this modality. Limitations of this study include the short duration of NIHFV, small sample size and lack of a control group. The only randomized trial evaluating this modality included 40 term infants with clinically diagnosed transient tachypnea of newborn (TTN) and concluded that the use of NIHFV leads to quicker recovery of TTN compared with the use of CPAP. However the assessment of recovery was subjective, and in a study that was unblinded could be ridden with bias. As well, many of those patients may not have required any form of NIV in the first place. Lastly a study by Czernik et al evaluated a group of 20 neonates at high risk of post-extubation failure who were prophylactically placed on NIHFV. Fourteen of the infants were successfully weaned off to NCPAP, but there was no control group to compare these results with. None of the four trials reported any adverse effects related to the use of NIHFV, although they were not powered to evaluate such outcomes.

At two of the investigators centres (Mount Sinai Hospital and the Hospital for Sick Children) NIHFV has been used as a rescue mode in recent months when NCPAP and/or BP-NCPAP has failed. In a review conducted [unpublished at this time] more than half the instances of its use (out of the 21 total cases) were due to increased spells (apneas, bradycardias and/or desaturations). In the six hours preceding and the six hours after initiation of NIHFV, the number of spells reduced from an average of 5.2 (±3.5) to 1.5 (±1.3). The majority of patients tried on NIHFV remained extubated, with less than a third eventually requiring re-intubation. As of yet, no reports of harm were directly linked with the use of NIHFV.

Despite limited evidence, NIHFV holds promise as an alternate mode of NIV. It may be superior to NCPAP/BP-NCPAP with respect to PaCO2 clearance from the lungs and also has the advantage of not requiring breath-synchronization, an issue that has hindered the widespread use of NIPPV. However, definitive assessment of the efficacy of NIHFV requires a prospective, randomized controlled trial. The goal of this study is to compare the rates of intubation when using BP-NCPAP vs. NIHFV as rescue mode of NIV post NCPAP failure in infants < 1,250 grams.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 72 hours post-natal age AND currently on NCPAP
* Less than 1,250 g when on NCPAP at time of enrollment

Exclusion Criteria:

* Congenital or acquired abnormality of upper airways
* Severe congenital anomalies including cyanotic congenital heart disease
* Severe nasal excoriation/injury preventing use of NIV interface
* Greater than 2,000 grams at time of randomization

Min Age: 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-06; Primary Completion 2014-11 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Failure of assignmed non-invasive mode post randomization to NIHFV or BP-CPAP | 72 hours

SECONDARY OUTCOMES:
Intubation rates at 72 hours and 7 days post randomization | 7 days
Comparison of the number of apneic spells | 7 days
PaCO2 levels at time of initiation | 2 hours
Total number of days on Endotracheal Mechanical Ventilation | 2 months
Rates of adverse outcomes between the 2 groups | 2 months
Time to discharge from hospital | 2 months
PaCO2 1 hour post NIV mode | 1 hour
Time to re-intubation | 7 days
Rates of intraventricular hemorrhage (IVH) | until discharge
Rates of BPD | until discharge

CONTACTS AND LOCATIONS:
Overall Officials: Vibhuti Shah, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Mukerji A, Sarmiento K, Lee B, Hassall K, Shah V. Non-invasive high-frequency ventilation versus bi-phasic continuous positive airway pressure (BP-CPAP) following CPAP failure in infants <1250 g: a pilot randomized controlled trial. J Perinatol. 2017 Jan;37(1):49-53. doi: 10.1038/jp.2016.172. Epub 2016 Sep 29. PMID 27684415